CLINICAL TRIAL: NCT03405285
Title: Clinical Evaluation of Connected Catheter Wireless Urinary Prosthesis for Management of Neurogenic Lower Urinary Tract Dysfunction
Brief Title: Connected Catheter Clinical Feasibility Study( CFS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Singularity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CoCath-01
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-07

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: Improved Bladder Management; Neurogenic Lower Urinary Tract Dysfunction; Bladder function following Spinal Cord Injury; Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connected Catheter Feasibility Study (Experimental): Clinical Feasibility Evaluation of Connected Catheter Wireless Urinary Prosthesis for Management of Neurogenic Lower Urinary Tract Dysfunction
  Interventions: Device: Connected Catheter

INTERVENTIONS:
Device: Connected Catheter — The Connected Catheter is a fully internal, urethral-indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization, including neurogenic lower urinary tract dysfunction (NLUTD - e.g. due to spinal cord injury). The CoCath is a sterile, single-extended-use device that resides fully internally to the male lower urinary tract (urethra + bladder neck) for an intended service life of up to 29 days per Catheter.

SUMMARY:
The objective of this study is to evaluate the safety and essential performance of the Connected Catheter System in males with neurogenic lower urinary tract dysfunction (NLUTD), both in an acute clinical setting, and during and extended period (up to 29 days) of home use.

DETAILED DESCRIPTION:
The Connected Catheter (C2P) is a replaceable urinary prosthesis that is intended for use in male patients 18 years of age or older who have impaired bladder emptying due to neurogenic lower urinary tract dysfunction, and who are capable of operating the device in accordance with the provided instructions for use, or who have trained caregivers capable of doing the same. The device must be replaced every 29 days

ELIGIBILITY:
Inclusion Criteria:

* Males age ≥ 18 with clinical diagnosis of neurogenic lower urinary tract dysfunction (NLUTD)
* Must be clinically suitable and capable of safely managing bladder using an intermittent voiding strategy Must have stable urinary management history with clean intermittent catheterization: no significant changes in bladder management regimen within past 12 months

OR:

Must have urodynamic profile suitable for CIC, as assessed via urodynamics study within past 12 months (including bladder capacity > 200mL without uninhibited bladder contractions)

* Subject's lower urinary tract anatomy (lengths of proximal and distal urethral must fall within the ranges serviceable by the Connected Catheter device, as specified in the investigational device instructions for use.
* For cases of NLUTD due to spinal cord injury, the subject must be in medically stable condition (i.e. post-spinal shock phase)

Exclusion Criteria:

* Active symptomatic urinary tract infection, as defined in this protocol (subjects may receive the CoCath Device after UTI has been treated)
* Significant risk profile or recent history of urethral stricture (e.g. stricture within past 90 days)
* Significant risk profile or recent history of clinically significant autonomic dysreflexia (e.g. History of hospitalization due to AD within past 12 months)
* Significant intermittent urinary incontinence (between catheterizations)
* Uninhibited bladder contractions and/or vesico-ureteral reflux that is not reliably controlled with medication or alternate therapy (e.g. botox injections)
* Pre-existing urinary pathologies and/or morphological abnormalities of the lower urinary tract or bladder (assessed during in-depth medical screening, including cystoscopy, urine analysis, and blood labs)
* Urinary tract inflammation or neoplasm
* Urinary fistula
* Bladder diverticulum (outpouching) > 5cm in size
* Chronic pyelonephritis (secondary to upper urinary tract infection(s) within past 6 months)
* Impaired kidney function or renal failure (assessed via blood creatinine levels > 2 mg/dL)
* Active gross hematuria
* Active urethritis
* Bladder stones
* Dependence on an electro-magnetic medical implant (e.g. cardiac pacemaker or implanted drug pump) or external device
* Individuals allergic or otherwise unable to take oral antibiotics
* Any physical or cognitive impairments that diminish the subject's ability to follow directions or otherwise safely use the CoCath System

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 5 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from genito-urinary injury/trauma | 29 Days
  Improved bladder management without injury or trauma to genito-urinary tract
Successful Acute Performance- I | On the day of Connected Catheter Insertion
  To evaluate successful retention of Connected Catheter and Void
Successful Acute Performance -II | On the day of Connected Catheter Insertion
  To evaluate successful bladder voiding with Connected Catheter
Successful Acute Performance- III | On the day of Connected Catheter Insertion
  To evaluate successful removal of Connected Catheter
Successful Acute Performance- IV | On the day of Connected Catheter Insertion
  To evaluate successful post-void sealing of Connected Catheter Valve
Successful Home-Use Performance | 29 days
  Successful Home-Use using same measures as Acute Performance

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - West Coast Urology, 11411 Brookshire Avenue, Suite 508, Downey, California
  - Tri Valley Urology, 25495 Medical Center Dr., Suite 204, Murrieta, California

IPD SHARING:
Plan to Share IPD: Undecided